CLINICAL TRIAL: NCT02179151
Title: Randomized, Double-Blind, Placebo Controlled, Phase 3 Trial of ZGN-440 (Subcutaneous Beloranib in Suspension) in Obese Subjects With Prader-Willi Syndrome to Evaluate Total Body Weight, Food-related Behavior, and Safety Over 6 Months
Brief Title: Double-Blind, Placebo Controlled, Phase 3 Trial of ZGN-440 (Beloranib) in Obese Subjects With Prader-Willi Syndrome
Acronym: bestPWS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: FDA Clinical Hold
Sponsor: Zafgen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZAF-311
Record Dates: First submitted 2014-06-25; First posted 2014-07-01 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Prader-Willi Syndrome; Obesity
Keywords: Prader-Willi Syndrome; Obesity; Hyperphagia
MeSH Terms: conditions — Prader-Willi Syndrome; Obesity; Hyperphagia | interventions — CKD732

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Intervention: ZGN-440 Placebo for Injectable Suspension
  Interventions: Drug: ZGN-440 Placebo for Injectable Suspension
- ZGN-440 Injectable Suspension (1.8 mg) (Experimental): Intervention: ZGN-440 for Injectable Suspension
  Interventions: Drug: ZGN-440 for Injectable Suspension
- ZGN-440 Injectable Suspension (2.4 mg) (Experimental): Intervention: ZGN-440 for Injectable Suspension
  Interventions: Drug: ZGN-440 for Injectable Suspension

INTERVENTIONS:
Drug: ZGN-440 for Injectable Suspension — Subjects will receive ZGN-440 twice weekly subcutaneous injections for up to 28 weeks.
  Other Names: ZGN-440; Beloranib
  Arms: ZGN-440 Injectable Suspension (1.8 mg); ZGN-440 Injectable Suspension (2.4 mg)
Drug: ZGN-440 Placebo for Injectable Suspension — Subjects will receive placebo twice weekly subcutaneous injections for up to 28 weeks.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of ZGN-440 (beloranib) in obese adolescent and adult subjects with Prader-Willi Syndrome.

DETAILED DESCRIPTION:
Phase 3, Randomized, Double-Blind, Placebo Controlled, Phase 3 Trial of ZGN-440 (Subcutaneous Beloranib in Suspension) in Obese Subjects with Prader-Willi Syndrome to Evaluate Total Body Weight, Food-related Behavior, and Safety Over 6 Months

ELIGIBILITY:
Inclusion Criteria:

* Confirmed genetic diagnosis of Prader-Willi Syndrome
* Age 12-65
* Obesity
* Age 12-17: BMI ≥ 95th percentile for age and gender
* Age 18-65: BMI ≥27 to ≤60 kg/m2

Exclusion Criteria:

* Subjects living in a group home ≥ 50% of the time
* Recent use (within 3 months) of weight loss agents including herbal medication
* Poorly controlled severe psychiatric disorders

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in total body weight | Baseline to Week 29
Change in hyperphagia-related behavior as measured by total score of a Hyperphagia Questionnaire | Baseline to Week 29

SECONDARY OUTCOMES:
Change in LDL cholesterol | Baseline to Week 29
Change in HDL cholesterol | Baseline to Week 29
Change in total body mass as measured by DXA | Baseline to Week 29
Change in total body fat mass as measured by DXA | Baseline to Week 29
Change in triglyceride | Baseline to Week 29

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Kim, MD, Study Director — Zafgen, Inc.
Locations (15):
- United States (15):
  - University of California, Davis, Sacramento, California
  - UCSD: Rady Children's Hospital, San Diego, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Kansas University Medical Center, Kansas City, Kansas
  - National Institute of Child Health, Bethesda, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - Children's Hospital and Clinics of Minnesota, Saint Paul, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Winthrop University, Mineola, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCandless SE, Yanovski JA, Miller J, Fu C, Bird LM, Salehi P, Chan CL, Stafford D, Abuzzahab MJ, Viskochil D, Barlow SE, Angulo M, Myers SE, Whitman BY, Styne D, Roof E, Dykens EM, Scheimann AO, Malloy J, Zhuang D, Taylor K, Hughes TE, Kim DD, Butler MG. Effects of MetAP2 inhibition on hyperphagia and body weight in Prader-Willi syndrome: A randomized, double-blind, placebo-controlled trial. Diabetes Obes Metab. 2017 Dec;19(12):1751-1761. doi: 10.1111/dom.13021. Epub 2017 Jul 13. PMID 28556449